CLINICAL TRIAL: NCT05249569
Title: Multi-center Phase II Open-label Study of Bavituximab, Axitinib, and Avelumab in Advanced Hepatocellular Carcinoma
Brief Title: Study of Bavituximab, Axitinib, and Avelumab in Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor pulled support for one of the study drugs.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, David Hsieh, Assistant Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0116
Record Dates: First submitted 2022-02-03; First posted 2022-02-21 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Axitinib; avelumab; bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axitinib / Avelumab /Bavituximab (Experimental): Axitinib 5 mg PO BID Avelumab 10 mg/kg IV every 2 weeks (2 doses in a 4-week cycle) Bavituximab 3 mg/kg IV every 1 week (4 doses in a 4-week cycle) Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.
  Interventions: Drug: Axitinib; Drug: Avelumab; Drug: Bavituximab

INTERVENTIONS:
Drug: Axitinib — Axitinib to be administered orally BID
Drug: Avelumab — Avelumab to be administered as a 1-hour IV infusion on Day 1 and Day 15 of each 28-day cycle.
Drug: Bavituximab — Bavituximab to be administered weekly on Days 1, 8, 15 and 22 of the 28-day cycle.

SUMMARY:
Across cancer types, immune checkpoint inhibitors have been shown to induce complete response, partial response, and stable disease after initial evidence of radiographic increase in tumor burden. Treatment beyond progression should be considered when the patient is stable (or improving) symptomatically and if tumor reassessment can be performed within a short period.

DETAILED DESCRIPTION:
Preclinical evidence indicates that VEGF and VEGF-dependent angiogenesis may induce immune suppression in tumors by impairing antigen presenting cells and effector T-cells, and enhancing T-regulatory cells and monocytes. Thus, targeting VEGF may reprogram the tumor immune microenvironment to render cancers more vulnerable to immunotherapies. Indeed, the use of anti-VEGF strategies as an immunotherapy adjuvant has been associated with clinical benefit in multiple cancer types including HCC, and no new safety signals. While the clinical benefit of monotherapy axitinib in HCC is modest, use of axitinib as an immunotherapy adjuvant may circumvent primary resistance mechanisms to immune checkpoint inhibitors in HCC leading to more frequent or robust anti-tumor immunity.

Given the complimentary immune augmenting mechanisms of targeting VEGF and phosphatidylserine, combination axitinib, bavituximab, and avelumab, a PD-L1 antibody, represents a novel and rational immunotherapy regimen in HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a histologically confirmed diagnosis consistent with HCC; known fibrolamellar HCC, or combined HCC-cholangiocarcinoma will be excluded.
2. Locally advanced or metastatic disease

   1. Patients with locally advanced or metastatic disease must have disease deemed not amenable to surgical and/or locoregional therapies or patients who have progressed following surgical and/or locoregional therapies.
   2. Measurable disease, as defined as lesions that can accurately be measured in at least one dimension according to RECIST version 1.1 at least 1 cm with contrast enhanced dynamic imaging (magnetic resonance imaging or computed tomography).
3. Availability of recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or slides (biopsied tumor lesion should not be a RECIST target lesion): 1) the biopsy or resection was performed within 2 years of AND 2) the patient has not received any intervening systemic anti-cancer treatment from the time the tissue was obtained.
4. Prior therapy is allowed provided the following are met: at least 4 weeks since prior locoregional therapy including surgical resection, chemoembolization, definitive radiotherapy with intent of disease control, or ablation. Provided target lesion has increased in size by 25% or more or the target lesion was not treated with locoregional therapy. Patients treated with palliative radiotherapy for symptoms will be eligible as long as the target lesion is not the treated lesion and radiotherapy will be completed at least 2 weeks prior to study drug administration.
5. Age ≥ 18 years
6. Child-Pugh Score A
7. ECOG Performance score of 0-1
8. Adequate organ and marrow function as defined below:

   1. Platelet count ≥ 50,000/mm3
   2. Hgb ≥ 8.5 g/dl
   3. Absolute neutrophil ≥ 1,500 cells/mm3
   4. Total bilirubin ≤ 2.0 mg/ml
   5. INR ≤ 1.7
   6. AST, ALT ≤5 times ULN
   7. Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
   8. albumin ≥ 2.5 g/dl
9. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) 4 weeks prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   a. A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
11. Subjects are eligible to enroll if they have non-viral-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

    1. HBV-HCC: Controlled (treated) hepatitis B subjects will be allowed if they meet the following criteria: Antiviral therapy for HBV must be given for at least 12 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. Subjects on active HBV therapy with viral loads under 100 IU/ml should stay on the same therapy throughout study treatment. Subjects who are anti-HBc (+), negative for HBsAg, negative for anti-HBs, and have an HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis.
    2. HCV-HCC: Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody. Patients who have failed HCV therapy as evidenced by detectable HCV RNA will be eligible. Subjects with chronic infection by HCV who are treated (successfully or treatment failure) or untreated are allowed on study. In addition, subjects with successful HCV treatment are allowed as long as there are ≥4 weeks between completion of HCV therapy and start of study drug. Successful HCV treatment definition: SVR12.
12. Ability to understand and the willingness to sign a written informed consent.
13. Patients who have received the vector, protein subunit, or nucleic acid COVID-19 vaccines are eligible to enroll.

Exclusion Criteria:

1. Prior liver transplant.
2. Prior systemic therapy directed at advanced or metastatic HCC.
3. Prior immunotherapy with IL-2, or anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
4. Prior therapy with axitinib or any prior therapies with other VEGF pathway inhibitors.
5. Clinically significant, uncontrolled heart disease and/or recent events including any of the following:

   1. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening).
   2. History of documented congestive heart failure (New York Heart Association functional classification III-IV).
   3. History of cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or pulmonary embolism within 6 months of screening.
   4. Patient has a left ventricular ejection fraction <40% as determined by MUGA scan or ECHO (MUGA and ECHO are not required prior to enrollment).
6. Known human immunodeficiency virus (HIV) positive (testing not required).
7. History of cerebrovascular accident, transient ischemic attack, or thromboembolic events (including both pulmonary embolism and deep venous thrombus but not including tumor thrombus) within the last 6 months.
8. Hypersensitivity to IV contrast; not suitable for pre-medication.
9. Active or fungal infections requiring systemic treatment within 7 days prior to screening.
10. Known history of, or any evidence of, interstitial lung disease or active noninfectious pneumonitis.
11. Evidence of poorly controlled hypertension which is defined as systolic blood pressure >159 mmHg or diastolic pressure >99 mmHg despite optimal medical management.
12. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
13. Active, known, or suspected autoimmune disease with the exception of subjects with vitiligo, type I diabetes mellitus, resolved childhood asthma or atopy. Subjects with suspected autoimmune thyroid disorders may be enrolled if they are currently euthyroid or with residual hypothyroidism requiring only hormone replacement. Subjects with psoriasis requiring systemic therapy must be excluded from enrollment.
14. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the study or compromise compliance with the protocol (e.g. chronic pancreatitis, active untreated or uncontrolled fungal, bacterial, or viral infections, etc.).
15. Known history of active bacillus tuberculosis.
16. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days of study administration. Inhaled or topical steroids and adrenal replacement doses >10 mg/day prednisone equivalents are permitted in the absence of autoimmune disease.
17. Patient who has received definitive radiotherapy with the sole intent of disease control ≤ 4 weeks prior to study entry. Palliative radiotherapy for symptomatic control (such as to bone metastases) is acceptable (if completed at least 2 weeks prior to study drug administration and no additional radiotherapy for the same lesion is planned).
18. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
19. Clinically apparent ascites on physical examination, ascites present on imaging studies is allowed.
20. Known severe hypersensitivity reactions to monoclonal antibodies (Grade 3).
21. Active gastrointestinal bleeding within previous 2 months.
22. History of any condition requiring anti-platelet therapy (aspirin >300 mg/day, clopidogrel >75 mg/day).
23. Diagnosis of any other malignancy within 5 years prior to screening visit, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, or low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (eg, surgery, radiation, or castration).
24. Prisoners or subjects who are involuntarily incarcerated.
25. History of leptomeningeal disease.
26. Symptomatic or clinically active brain metastases.
27. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after contraception and until the termination of gestation, confirmed by a positive hCG laboratory test.
28. Has dual active HBV infection (HBsAg (+) and /or detectable HBV DNA) and HCV infection (anti-HCV Ab(+) and detectable HCV RNA) at study entry.
29. Known prior or suspected hypersensitivity to study drugs or any component in their formulations.
30. Current use or anticipated need for drugs that are known strong CYP3A4/5 inducers, including their administration within 10 days prior to patient receiving the first study treatment, eg, phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St John's wort.
31. Patients with 2+ proteinuria on urine dipstick analysis and confirmed to have ≥2 grams of protein in a 24-hour urine collection.
32. Current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors, including their administration within 10 days prior to patient receiving the first study treatment, (eg, grapefruit juice or grapefruit/grapefruit-related citrus fruits, ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hsieh, MD, Principal Investigator — Assistant Professor
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axitinib / Avelumab /Bavituximab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Sponsor pulled support for one of the study drugs. | 1

BASELINE CHARACTERISTICS:
Population: One patient signed consent and was enrolled on study. However, the sponsor that was planning to provide one of the study drugs decided they no longer wanted to supply the drug for this project. The participant that was enrolled on the study did not receive treatment before the study was terminated.
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Combination Therapy
Description: To determine the objective response rate of combination axitinib,avelumab, and bavituximab in advanced HCC not previously treated with systemic therapy.
Time Frame: Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months.
Population: One patient signed consent and was enrolled on study. The participant that was enrolled on the study did not receive treatment before the study was terminated. Data was not collected for this outcome measure.
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease Control Rate
Description: To determine the disease control rate of response of combination axitinib, bavituximab, and avelumab compared to historical controls.
Time Frame: Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 48 months.
Population: as for outcome 1
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: To determine the overall survival, 6 of combination axitinib, bavituximab, and avelumab compared to historical controls.
Time Frame: as for outcome 2
Population: as for outcome 1
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

4. Secondary Outcome: 6-month Progression-free Survival
Description: To determine the 6-month progression-free survival of combination axitinib, bavituximab, and avelumab compared to historical controls.
Time Frame: as for outcome 2
Population: as for outcome 1
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Description: To determine the duration of response of combination axitinib, bavituximab, and avelumab compared to historical controls.
Time Frame: as for outcome 2
Population: as for outcome 1
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Safety Profile as Measured by the Number of Participants With AEs (Serious / Non-serious) as Graded by NCI CTCAE v5.0
Description: Safety profile of combination axitinib, bavituximab, and avelumab will be measured by the number of participants with Adverse Events (AEs) (serious / non-serious) as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: as for outcome 2
Population: as for outcome 1
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

7. Secondary Outcome: Safety Profile as Measured by the Number of Participants With Lab Abnormalities as Graded by NCI CTCAE v5.0
Description: Safety profile of combination axitinib, bavituximab, and avelumab will be measured by the number of participants with lab abnormalities as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: as for outcome 2
Population: One patient signed consent and was enrolled on study.The participant that was enrolled on the study did not receive treatment before the study was terminated. Data was not collected for this outcome measure.
Arm/Group | Axitinib / Avelumab /Bavituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Axitinib / Avelumab /Bavituximab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT05249569/Prot_SAP_000.pdf